CLINICAL TRIAL: NCT03413280
Title: The Effectiveness of Preemptive Effect of Rectus Sheath Block and Intercostal Block on Postoperative Visceral Pain in Laparoscopic Cholecystectomy
Brief Title: Preemptive Analgesic Effects of Rectus Sheath Block in Laparoscopic Cholecystectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hyuk Lee, clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017-0301
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Preemptive Peripheral Nerve Block; Pain, Postoperative; Acute Pain
Keywords: preemptive analgic effect; Rectus Sheath Block; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative Rectus sheath block: group Pre (Experimental): ultrasound guided Rectus sheath block block with 0.25% ropivacaine 40ml Before surgical incision
  Interventions: Drug: Ultrasound guided Rectus sheath block; Drug: Intercostal nerve block
- postoperative Rectus sheath block: group Post (Active Comparator): ultrasound guided Rectus sheath block block with 0.25% ropivacaine 40ml After surgical incision
  Interventions: Drug: Ultrasound guided Rectus sheath block; Drug: Intercostal nerve block

INTERVENTIONS:
Drug: Ultrasound guided Rectus sheath block — Ultrasound guided rectus sheath block with 0.25% ropivacaine 34ml around umbilicus
Drug: Intercostal nerve block — Ultrasound guided intercostal nerve block with 0.25% ropivacaine 6ml in 7,8,9 th intercostal space

SUMMARY:
The purpose of this study was to investigate the effectiveness of preemptive effect of rectus sheath block (RSB) and intercostal nerve block (ICNB) on postoperative visceral pain in laparoscopic cholecystectomy (LLC).

After induction of general anesthesia, group of patient is decided randomly. In Group pre, RSB and ICNB are performed with 0.25% Ropivacaine 40ml before the operation. In Group post, RSB and ICNB are performed with 0.25% Ropivacaine 40ml after the operation.

Measure the NRS and compare the rescue analgesic dose used at 0, 0.5, 1, 2, 6, 9, 18, and 24 hours after arrival at the recovery room.

ELIGIBILITY:
Inclusion Criteria:

1. adults between the ages of 20 and 80
2. scheduled laparoscopic cholecystectomy patient
3. ASA class 1 or 2
4. Patients who have voluntarily agreed in writing to participate in the trial

Exclusion Criteria:

1. Patient with side effects on local anesthetics or steroids
2. Patient who are taboo of peripheral nerve block such as blood clotting disorder, infection, etc.
3. Patients with uncontrolled medical or psychiatric problem
4. Patient does not agree to participate in the study
5. Patients who are pregnant or lactating
6. Patients whose visceral pain is expected to be too severe
7. Patients receiving a single laparoscopic cholecystectomy (including using a robot)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Difference of analgesic consumption between both group | at 0, 0.5, 1, 2, 6, 9, 18, 24 hours after operation
  The difference in analgesics usage between the two groups after the operation is checked at fixed intervals (at 0, 0.5, 1, 2, 6, 9, 18, 24 hours after operation) to compare.

SECONDARY OUTCOMES:
compare the Numeric rating scale (NRS) | at 0, 0.5, 1, 2, 6, 9, 18, 24 hours after operation
  The Numeric Rating Scale (NRS-11) is an 11-point scale for patient self-reporting of pain. It is for adults and children 10 years old or older.
  0: No pain, 1-3: mild pain, 4-6: Moderate pain, 7-10: severe pain, 10: worst pain imaginable.
  After surgery, the NRS differences between the two groups were compared at a constant interval (0, 0.5, 1, 2, 6, 9, 18, 24 hours postoperatively).

CONTACTS AND LOCATIONS:
Overall Officials: JongHyuk Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea